CLINICAL TRIAL: NCT01536132
Title: Multicenter, Double-blind, Placebo-controlled Randomized Trial to Evaluate the Efficacy and Safety of Intravenous Administration of Intermittent Doses of Levosimendan in Ambulatory Patients With Advanced CHF: the LION-HEART Study
Brief Title: Intermittent Intravenous Levosimendan in Ambulatory Advanced Chronic Heart Failure Patients
Acronym: LION-HEART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Josep Comín, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMIM-LEV-0901
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: Levosimendan; chronic heart failure; inotropic drug
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosimendan (Active Comparator): levosimendan at a dose of 0.2 micrograms/kg/min for 6 hours intravenous infusion
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): placebo (same appereance than levosimendan in colour) at a dose of 0.2 micrograms/kg/min for 6 hours intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — 0.2 micrograms/kg/min is administered intravenously without bolus for 6 hours every two weeks.
  Other Names: SIMDAX (trade mark)
  Arms: Levosimendan
Drug: Placebo — Placebo (same appearance than active drug) is administered with the same dosing regime
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of intravenous administration of intermittent doses of levosimendan (infusions of 0,2 μg/kg/min, of levosimendan or placebo, without bolus, for 6 hours every 2 weeks) compared to placebo in ambulatory patients with advanced chronic heart failure.

DETAILED DESCRIPTION:
The LION-HEART study (Levosimendan® Intermittent administration in Outpatients: effects on Natriuretic peptides in advanced chronic HEART failure) was a multicenter, double-blind, randomized, parallel group, placebo-controlled trial evaluating the efficacy and safety of intravenous administration of intermittent doses of levosimendan in outpatients with advanced chronic heart failure.

Study Design and Oversight Between November 2010 and December 2012,69 patients fulfilling inclusion criteria were enrolled from 12 recruiting centers in Spain (Figure 1). The study protocol was approved by institutional review board of each participating center and conducted in accordance with the principles of the Declaration of Helsinki (1996), International Conference on Harmonization Good Clinical Practice, and local and national regulations. All enrolled patients provided written informed consentbefore any study-related procedure was undertaken. The study was registered on the website www.ClinicalTrials.gov (unique identifier: NCT01536132) and the EudraCT database (2009-014242-28). The trial was designed, implemented and overseen by the Steering Committee. On-site monitoring of the study, data collection and data management was performed by a Clinical Research Organization (CRO, 3DHealth). The manuscript was written and submitted by the Steering Committee members. All contributing authors had full access to study data and analyses.

Study population, eligibility and recruitment The study was divided in three different parts: 1) screening (1 week), 2) treatment (12 weeks) and 3) follow-up (12 weeks). An additional vital status assessment was planned after 12 months of enrolment (Figure 2, design of the study).

Eligibility was assessed at the screening phase, once the written informed consent was obtained. Inclusion criteria for this study were: age over 18 years, left ventricular ejection fraction (LVEF) of less than 35% measured in the previous 6 months and clinical diagnosis of advanced chronic HF (Metra M et al. Eur J Heart Fail 2007; 9(6-7):684-694)according to the following criteria: a) presence for >3 months of typical signs and symptoms of HF b) persistent ambulatory NYHA functional class III or IV for the last 4 weeks, c) no signs of congestion or low cardiac output at the time of enrolment, d) episodes of pulmonary and/or systemic congestion requiring intravenous administration of diuretics (either hospitalized or in an ambulatory basis) in the previous 12 months, e) all the previous criteria were present despite optimal medical management (including use of diuretics, antagonists of the renin-angiotensin-aldosterone system and beta-blockers) and device therapy (including implantable cardioverter defibrillator-ICD and/or cardiac resynchronization therapy-CRT) or attempts to optimize it. Major exclusion criteria were: concurrent inclusion in another study, the presence of left ventricular tract obstruction, uncorrected significant primary valve disease, recent acute coronary syndrome or stroke, hypertrophic or restrictive cardiomyopathy, administration of amrinone, milrinone, enoximone, dopamine or dobutamine in the previous 3 days, administration of levosimendan in the previous 31 days, serum potassium below 3.5mmol/L, estimated glomerular filtration rate <30ml/min/m2 (MDRD-4 formula), systolic blood pressure < 90 mmHg orheart rate > 110 bpm at screening, planned or ongoing evaluation for any of the following procedures: CRT, ICD, coronary revascularization, heart transplant or left ventricular assist device (LVAD) implant, other acute or chronic conditions that would made the patient unsuitable for this study according to the investigator's judgement, anticipated poor compliance and inability or unwillingness to give informed consent.

Randomization and Blinding Eligible patients that signed the informed consent were randomized in a 2:1 ratio to receive either Levosimendan or placebo. Randomization was centrally conducted and supervised by the CRO. The computer-generated randomization scheme used random permuted blocks stratified per center. Once the patient was allocated to Levosimendan of placebo, the CRO communicated the exact treatment number to the local hospital pharmacy which handed out the treatment to the local investigator at each infusion cycle. Levosimendan and placebo had the same appearance thus the treatment was concealed to both investigators and study patients (double blind).

Therapy Patients were randomized in a 2:1 ratio to receive either Levosimendan or placebo (i.e. two patients assigned Levosimendan for every one patient assigned placebo) as an intermittent dosing (every two weeks) by a 6-hour intravenous infusion (0.2 μg / kg / min without bolus) for a period of 12 weeks (6 cycles) in study patients with advanced chronic heart failure.In case of hypotension (systolic blood pressure <90 mmHg or <100 mmHg with symptoms) or clinical intolerance to the drug, the dose could be reduced to 0.01 μg /kg/min. Furtherreduction to 0.05μg/kg/min or discontinuation of the drug waspossible if these adverse effects persisted.Study treatment was administered during a maximum of 12 weeks in an ambulatory administration setting that allowed non-invasive monitoring of vital signs. During the first infusion, 24-hour ECG monitoring (either with ambulatory Holter monitoring or telemetry) was required for safety evaluations.

After the treatment period, patients were followed every 4 weeks for 12 additional weeks. At the end of the study, patients were followed for a maximum of 12 months - i.e. the last visit (vital status assessment)was performed 9 months after the last administration of study treatment.

Data collection Baseline information was obtained in stable patients without signs of fluid overload or low-cardiac output after written informed consent. These data included medical history, hospitalizations, relevant clinical and demographic information and physical examination by means of direct interview, examination and medical record review and included NYHA class, most recent LVEF, medical therapy and 12-lead ECG. These data, including the occurrence of adverse events and hospitalizations was re-evaluated every two weeks the first 3 months and every 4 weeks the next 3 months. Additional evaluations at baseline included self-assessment of patient reported outcomes (PRO, including health-related quality of life-HR-QoL- evaluated by means of the generic EQ-5D and the HF specific Kansas City Cardiomyopathy Questionnaire, KCCQ), local laboratory measurements, and the distance walked in the 6 minutes walking test (6MWT). PRO and 6 MWT were re-evaluated at week 13 and week 25. Vital status assessment was also performed after 12 months of inclusion into the study. Measurements of serum amino-terminal B-type pro-natriuretic peptide (NT-proBNP, pg/mL) were performed locally with and immunoassay based on chemiluminescence using the Elecsys System (Roche®) before and 24 h after initiation of each study drug infusion (either Levosimendan or placebo).

Follow-up and Evaluation of end-points The primary end-point of efficacy in the LION-HEART study was to determine, relative to placebo, the effect of 6 cycles of ambulatory 6-hour intravenous infusions of levosimendan every two weeks on concentrations of NT-proBNP throughout the 12-week treatment period in patients with advanced chronic heart failure.

Secondary End-points of safety and efficacy The secondary objectives for efficacy included the evaluation of the effect of the drug compared to placebo on functional variables including NYHA class, patient centered outcomes including HR-QoL, the relative change in values of NT-proBNP from baseline to the end of treatment and unplanned hospitalizations (for HF, for cardiovascular reasons and all-cause). As additional pre-specified efficacy end-points the report of combined all-cause death or other terminal events (urgent LVAD or heart transplant) with hospitalization was planned. The safety objectives aimed to evaluate the effect of the study drug compared to placebo on all-cause mortality, changes in renal and liver function. The impact of the administration of the study drug on heart rate and the risk of development of life-threatening arrhythmias were investigated in all patients in our study.

All adverse events, serious and non-serious were prospectively evaluated and recorded. Data safety was regularly reviewed by medical personnel of the CRO without any contact with investigators or patients on an ongoing basis according to the qualification of major events (death, readmission) and other adverse events. Since allocation of patients to the study drug or placebo was concealed, adjudication of adverse events and secondary efficacy end-points(including death and hospitalizations) was undertaken by each local principal investigator at each recruiting center.

For efficacy, safety and tolerability evaluations, an intention to treat analysis was undertaken in all patients that received at least one study drug infusion. Adverse events are reported following the Medical Dictionary for Regulatory Activities (MeDRA) definitions.

ELIGIBILITY:
Inclusion Criteria:

* qged more than 18,
* left ventricular ejection fraction below 35%,
* diagnostic criteria of advanced chronic heart failure.

Exclusion Criteria:

* Conduction abnormalities (auricular ventricular block),
* malignant arrythmias,
* recent administration of inotropic drugs,
* recent acute coronary syndrome,
* recent cerebrovascular accident,
* glomerular filtration rate below 30,
* systolic blood pressure below 90 mmhg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes of natriuretic peptide levels between baseline and end of treatment. | 3 months.

SECONDARY OUTCOMES:
Mortality . | from baseline to end of follow-up (12 months).
Hospitalisation. | from baseline to end of follow-up (12 months).

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP COMIN COLET, MD PHD, Study Chair — HOSPITAL DEL MAR MEDICAL RESEARCH INSTITUTE
Locations (13):
- Spain (13):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Valdecillas, Santander, Cantabria
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Virgen de la Victoria, Málaga, Malaga
  - Hospistal Central Asturias, Oviedo, Principality of Asturias
  - Complexo Hospitalario A Coruña, A Coruña, Spain
  - Hospital Virgen Arrixaca, Murcia, Spain
  - Hospital Virgen del Rocío, Seville, Spain
  - Hospital la Fe, Valencia, Spain
  - Hospital Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No